CLINICAL TRIAL: NCT04435834
Title: Cerebral Hemodynamics- ICHOR II
Brief Title: Individual Cerebral Hemodynamic Oxygenation Relationships
Acronym: ICHOR
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Matthew Borzage (Other)
Responsible Party: Sponsor-Investigator, Matthew Borzage, Principal Investigator, Children's Hospital Los Angeles
Organization: Children's Hospital Los Angeles (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: CHLA-20-00136
Record Dates: First submitted 2020-06-10; First posted 2020-06-17 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Anesthesia; Anesthesia; Reaction
Keywords: Magnetic Resonance Imaging; Cerebral Blood Flow; Cerebral Metabolism; Anesthesia
MeSH Terms: interventions — Propofol; Sevoflurane

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized in a stratified, blocked study design. Stratification is based on two factors: gestational age (2 groups: ≥37 weeks and ≤37 weeks) and postmenstrual age at MRI (2 groups: ≥37 weeks and ≤37 weeks). Blocking of each stratum is performed in groups of 4.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Participant and care provider will be aware randomization status. Investigator and outcomes assessor will be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Propofol (Experimental): Subject will receive propofol anesthesia during their MRI. Dosage form: injectable solution. Dosage: 100-300 mcg/kg/min, or as per clinical standard of care appropriate for specific subjects.
  Frequency and duration: continuous infusion while undergoing MRI.
  Interventions: Drug: Propofol or Sevoflurane
- Sevoflurane (Experimental): Subject will receive sevoflurane anesthesia during their MRI. Dosage form: volatile liquid for inhalation Dosing: 0-1 month full term neonate (3.3% in oxygen), 1-6 months old (3% in oxygen), 6 months to <3 years old (2.8% in oxygen), or as per clinical standard of care appropriate for specific subjects.
  Frequency and duration: continuous infusion while undergoing MRI.
  Interventions: Drug: Propofol or Sevoflurane

INTERVENTIONS:
Drug: Propofol or Sevoflurane — Patient's will be randomized to the group receiving propofol, or the group receiving sevoflurane.

SUMMARY:
This is a randomized controlled trial in patients who require clinical anesthesia. The main purpose of this study is to understand whether there are differences in the cerebral blood flow, and oxygen metabolism affected by two types of anesthesia: propofol or sevoflurane. Subjects who require clinical anesthesia for a clinical MRI and for whom the use of propofol and sevoflurane are in clinical equipoise will be offered to have the anesthesia they will receive during their MRI randomized. All eligible subjects will be asked to provide informed consent before participating in the study.

DETAILED DESCRIPTION:
This is a randomized controlled trial in patients who require clinical anesthesia. The main purpose of this study is to understand whether there are differences in the cerebral blood flow, and oxygen metabolism affected by two types of anesthesia: propofol or sevoflurane. Subjects who require clinical anesthesia for a clinical MRI and for whom the use of propofol and sevoflurane are in clinical equipoise will be offered to have the anesthesia they will receive during their MRI randomized. All eligible subjects will be asked to provide informed consent before participating in the study.

Treatment:

All patients will be screened to ensure propofol and sevoflurane are in clinical equipoise. Those who meet eligibility criteria, and who undergo the informed consent, will be randomize to receive propofol or sevoflurane during their MRI. Standard-of-care anesthesia safety, dose and monitoring will not be changed. During their MRI, additional images will be acquired that measure the cerebral blood flow and cerebral venous oxygenation. These additional images will take up-to 10 extra minutes to acquire. This will increase the duration each subject spends under anesthesia, and in the MRI scanner by up-to a total of 10 extra minutes.

Safety Assessment:

To ensure that either propofol or sevoflurane are in clinical equipoise, all patients will be screened by an anesthesiologist. The experiment will occur in the standard-of-care clinical MRI environment. All patient safety and monitoring will remain in place. Throughout the induction, maintenance and recovery from anesthesia, all procedures will occur in the standard of care environment and will be overseen by trained clinical personnel.

Efficacy Assessment:

Cerebral blood flow and metabolism MRIs will be collected from all subjects.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are scheduled for a clinically indicated MRI at the sponsor institution.
* Patients who are able to tolerate an MRI.
* Patients who require clinical anesthesia for their MRI.
* Patients with conditions not believed to alter oxygen metabolism or blood flow in the brain, including but not limited to patients with orthopedic indications, undescended testicles, hernia repairs, term equivalent age scans.
* Patients who have no medical conditions that make the use of propofol or sevoflurane better for their clinical outcome.
* Patients between birth and up-to 1 year of age.
* Patients with conditions known to alter oxygen metabolism or blood flow in the brain, e.g. traumatic brain injury, hypoxic ischemic encephalopathy, tumor.

Exclusion Criteria:

* Patients with an MRI-incompatible device or implant (e.g. pacemakers, stents)
* Preterm infants less than 25 weeks postmenstrual age (PMA) at the time of the scan.
* Patients who are clinically too unstable to extend their MRI by up-to 10 minutes.
* Patients who do not require clinical anesthesia.
* Patients at risk for propofol infusion syndrome (known severe metabolic acidosis, hyperkalemia, lipemia, rhabdomyolysis, hepatomegaly, renal failure, ECG ST segment elevation, and/or cardiac failure)
* Patients at risk for sevoflurane-based malignant hyperthermia (known ryanodine receptor mutations)
* Patient at risk for sensitivity to volatile halogenated anesthetic agents (known congenital Long QT Syndrome or patients taking drugs that can prolong the QT interval),
* Patients with Perioperative Hyperkalemia (known neuromuscular disease, particularly Duchenne muscular dystrophy)

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2020-06-09 (Actual); Primary Completion 2026-09-10 (Estimated); Study Completion 2026-09-10 (Estimated)

PRIMARY OUTCOMES:
Change in cerebral blood flow (ml blood/100g/min) | Time points over which the change is assessed: change from (1) start of MRI, through (2) MRI completion, an average of 60 minutes.
  Phase contrast (PC) acquisition via MRI will be used to assess any impact of anesthesia on cerebral blood flow.
Change in cerebral metabolic rate of oxygen (ml O2/100g/min) | Time points over which the change is assessed: change from (1) start of MRI, through (2) MRI completion, an average of 60 minutes.
  T2 relaxation under spin tagging (TRUST) acquisition via MRI will be used to assess any impact of anesthesia on cerebral metabolic rate of oxygen.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Borzage, PhD, Principal Investigator — Children's Hospital Los Angeles
Locations (1):
- Children's Hospital Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No